CLINICAL TRIAL: NCT07234214
Title: Comparison of Five Osteotomy Protocols on Implant Stability and Patient Anxiety: A Randomized Controlled Clinical Trial
Brief Title: Randomized Trial of Five Implant Osteotomy Protocols on Stability and Anxiety
Acronym: OSTEO-ISQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sercan Küçükkurt (Other)
Responsible Party: Sponsor-Investigator, Sercan Küçükkurt, Associate Professor, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IAU-OMS-OSTEO-RCT-01; IAU Ethics Approval 2023/141 (Other: Istanbul Aydın University Institutional Review Board)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant Surgery; Osteotomy Protocols
Keywords: Dental implants; Osteotomy protocols; Implant stability; Insertion torque; Resonance frequency analysis; Osseodensification; Bone condensation; Patient anxiety

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, parallel-group clinical trial comparing five different implant osteotomy techniques with respect to insertion torque, implant stability, and patient-reported anxiety.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The surgeon could not be blinded due to the nature of the interventions. However, implant stability was measured by an independent assessor, and statistical analyses were performed by a blinded biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 50 rpm - Ultra-low-speed drilling (Experimental): Sequential osteotomy drilling at 50 rpm without irrigation, followed by implant placement.
  Interventions: Procedure: Osteotomy technique - 50 Rpm
- 300 rpm - Moderate-speed drilling (Experimental): Sequential osteotomy drilling at 300 rpm with external irrigation, followed by implant placement.
  Interventions: Procedure: Osteotomy technique - 300 Rpm
- 800 Rpm - High-speed drilling (Experimental): Sequential osteotomy drilling at 800 rpm with external irrigation, followed by implant placement.
  Interventions: Procedure: Osteotomy technique - 800 Rpm
- DNS - Osseodensification (Experimental): Osteotomy prepared with Densah® burs (Versah, USA) at 1200 rpm counterclockwise with irrigation, following pilot drilling.
  Interventions: Procedure: Osteotomy technique - DNS (Osseodensification)
- CDS - Bone condensation (Experimental): Osteotomy prepared with condenser drills (Surgident, South Korea) at 50 rpm clockwise without irrigation, following pilot drilling at 800 rpm.
  Interventions: Procedure: Osteotomy technique - CDS (Bone Condensation)

INTERVENTIONS:
Procedure: Osteotomy technique - 50 Rpm — Ultra-low-speed sequential drilling at 50 rpm without irrigation.
  Arms: 50 rpm - Ultra-low-speed drilling
Procedure: Osteotomy technique - 300 Rpm — Moderate-speed sequential drilling at 300 rpm with irrigation.
  Arms: 300 rpm - Moderate-speed drilling
Procedure: Osteotomy technique - 800 Rpm — High-speed sequential drilling at 800 rpm with irrigation.
  Arms: 800 Rpm - High-speed drilling
Procedure: Osteotomy technique - DNS (Osseodensification) — Osseodensification using Densah® burs at 1200 rpm counterclockwise with irrigation.
  Arms: DNS - Osseodensification
Procedure: Osteotomy technique - CDS (Bone Condensation) — Bone condensation with condenser drills at 50 rpm clockwise without irrigation.
  Arms: CDS - Bone condensation

SUMMARY:
This clinical trial is studying different methods of preparing bone for dental implants. When a tooth is missing, a small titanium screw called a dental implant can be placed in the jaw to replace it. The stability of the implant during the first weeks after surgery is very important for long-term success.

In this study, 100 patients each received a single dental implant. They were randomly assigned to one of five surgical methods: drilling at 50, 300, or 800 revolutions per minute (rpm), bone densification using special burs, or bone condensation using condenser drills. The goal was to compare how these techniques affect implant stability, measured by insertion torque and resonance frequency analysis, as well as the patient's anxiety before and after surgery.

This research aims to find which technique provides the best balance between bone healing and patient comfort. All participants were healthy adults, and the study was approved by the institutional ethics committee.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial was conducted at Istanbul Aydın University, Department of Oral and Maxillofacial Surgery, between 2019 and 2023. A total of 100 systemically healthy adults requiring a single dental implant in a healed edentulous ridge were enrolled. Patients were randomly assigned (n = 20 per group) to one of five osteotomy protocols:

Sequential drilling at 50 rpm without irrigation

Sequential drilling at 300 rpm with irrigation

Sequential drilling at 800 rpm with irrigation

Osseodensification with densifying burs at 1200 rpm (counterclockwise, irrigated)

Bone condensation using condenser drills at 50 rpm (clockwise, non-irrigated, following pilot drilling)

The same tapered titanium implant system was used in all patients. Primary outcomes were insertion torque (Ncm) and implant stability quotient (ISQ) measured at placement and at 1 week, 1 month, 2 months, and 3 months. The secondary outcome was patient-reported anxiety assessed on a visual analog scale (VAS) pre- and postoperatively.

Bone density was evaluated preoperatively using cone-beam computed tomography (CBCT, expressed as Hounsfield Unit Equivalents) and intraoperatively classified by Misch criteria. Patients with insertion torque < 25 Ncm were excluded from stability analysis and allowed to heal submerged.

The trial followed the CONSORT statement and adhered to the Declaration of Helsinki. Ethical approval was obtained (IAU 2023/141). Results are expected to clarify whether moderate-speed drilling, high-speed drilling, ultra-low-speed drilling, or non-subtractive approaches (osseodensification, condensation) provide the most favorable outcomes in terms of implant stability and patient psychological response.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-78 years
* Single-tooth healed edentulous ridge
* First-time implant candidates
* Preoperative cone-beam computed tomography (CBCT) available
* American Society of Anesthesiologists (ASA) Physical Status I
* Non-smokers or light smokers (<10 cigarettes/day)
* Provided written informed consent

Exclusion Criteria:

* Previous grafting or sinus augmentation at the implant site, including socket grafting after extraction
* Systemic contraindications to implant surgery
* Intraoperative complications or postoperative infections
* Missing insertion torque (IT) or ISQ data
* Requirement for a submerged (two-stage) protocol
* Deviations from the standardized surgical protocol or implant system

Ages: 20 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Insertion Torque at Implant Placement | At the time of implant placement.
  Maximum insertion torque (Ncm) recorded at implant placement using a calibrated surgical motor and confirmed with a manual torque wrench when needed.
Implant Stability Quotient (ISQ) | At baseline, 1 week, 1 month, 2 months, and 3 months after implant placement.
  Implant stability measured by resonance frequency analysis (RFA) using the Osstell Mentor™ device. Mean of buccolingual and mesiodistal measurements recorded.

SECONDARY OUTCOMES:
Change in Patient-Reported Anxiety (VAS) | Preoperative (within 30 minutes before surgery) and immediate postoperative (within 30 minutes after surgery).
  Visual analog scale (0-10; 0 = no fear, 10 = extreme fear). Difference between preoperative and immediate postoperative scores.
Procedure-Related Adverse Events | From surgery to 3 months.
  Number of participants with any procedure-related adverse event (e.g., postoperative infection, sensory disturbance, early implant failure requiring removal, wound dehiscence). Events assessed clinically and recorded at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konuklu R, Kucukkurt S. Comparison of Five Osteotomy Protocols on Implant Stability and Postoperative Anxiety: A Randomized Controlled Trial. Clin Implant Dent Relat Res. 2026 Feb;28(1):e70125. doi: 10.1111/cid.70125. PMID 41664595